CLINICAL TRIAL: NCT07290049
Title: Evaluation of Postoperative Pain After Pulpotomy Using Calcium Silicate Cements in Permanent Molars With and Without Laser Biomodulation: A Randomized Clinical Trial
Brief Title: Postoperative Pain After Pulpotomy in Children Using Calcium Silicate Cements With and Without Laser Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fujairah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UOF REC2025-04-22
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Irreversible Pulpitis; Symptomatic Irreversible Pulpitis (SIP)
Keywords: Vital Pulp Therapy; Pulpotomy; Irreversible Pulpitis; Postoperative Pain; Calcium Silicate Cement; Bioceramic; Laser Biomodulation; Er,Cr:YSGG Laser; EndoCem; Biodentine; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group study. Participants are randomly assigned to one of two intervention groups and remain in that group for the entirety of the study. The groups are treated concurrently, and their outcomes are compared directly to each other.
  Group 1 (Control): Receives the standard pulpotomy procedure using the calcium silicate cement (EndoCem).
  Group 2 (Intervention): Receives the standard pulpotomy procedure with the addition of laser biomodulation prior to the placement of the calcium silicate cement (EndoCem).
  There is no crossover or sequential assignment of interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The operating clinician performing the pulpotomy procedure cannot be blinded due to the nature of the laser intervention. However, to maintain blinding, this clinician will not be involved in postoperative assessments. The participant, the independent assessor who collects the pain scores (Outcomes Assessor), and the statistician analyzing the final data will all be unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoCem Pulpotomy (Active Comparator): Participants in this arm will receive a full pulpotomy procedure for the treatment of symptomatic irreversible pulpitis. Following coronal pulp removal and hemostasis, the vital radicular pulp tissue will be covered with the calcium silicate cement EndoCem (ZTM Medicare, Pre-mixed MTA Putty), applied according to the manufacturer's instructions. The tooth will then receive a final restoration. This arm serves as the active comparator, evaluating the standard vital pulp therapy protocol using a modern bioceramic material.
  Interventions: Device: Calcium Silicate Cement
- EndoCem + Laser Pulpotomy (Experimental): Participants in this arm will receive an identical full pulpotomy procedure. However, prior to the placement of the EndoCem cement, the exposed radicular pulp stumps will undergo Er,Cr:YSGG laser biomodulation. The laser will be applied in a non-ablative, biostimulatory mode using specific parameters (e.g., 1.0 W, 20 Hz, 50 mJ, 60% water, 70% air) for a predetermined duration to achieve the biomodulation effect. Following laser application, EndoCem cement is placed and the tooth is restored. This is the experimental arm investigating the adjunctive effect of laser therapy.
  Interventions: Device: Calcium Silicate Cement; Device: Er,Cr:YSGG Laser

INTERVENTIONS:
Device: Calcium Silicate Cement — A premixed, ready-to-use hydraulic tricalcium silicate cement (commercial name: EndoCem MTA Pre-mixed Putty) used as a direct pulp-capping agent. It is applied over the vital radicular pulp tissue following a pulpotomy procedure to seal the pulp chamber and promote healing and reparative dentin formation. The material is used according to the manufacturer's instructions for vital pulp therapy.
Device: Er,Cr:YSGG Laser — An Erbium, Chromium: Yttrium-Scandium-Gallium-Garnet laser system used in a non-ablative, low-level power setting for biomodulation. Following hemostasis in the pulpotomy procedure, the laser tip delivers photonic energy to the exposed pulp stumps in a defocused, non-contact mode. The intended biological effects are biostimulation of pulpal cells, enhanced healing, and anti-inflammatory action, which may reduce postoperative pain. Specific parameters (e.g., power, frequency, air/water coolant ratio) are set for therapeutic bio-stimulation rather than surgical cutting.
  Arms: EndoCem + Laser Pulpotomy

SUMMARY:
This study is for children and young adults who have a severe toothache in a permanent back molar, caused by an inflamed nerve (a condition called irreversible pulpitis). Usually, the treatment for this is a root canal, which removes the entire nerve. However, a different treatment called "vital pulp therapy" or "pulpotomy" may be an option. This simpler procedure removes only the infected part of the nerve, leaving the healthy part alive, and then seals the tooth with a special material.

The goal of our research is to see if we can make this pulpotomy procedure even more comfortable for patients afterward. We are testing two approaches:

Using a modern dental filling material called EndoCem to seal the tooth.

Using the same EndoCem material, but first applying a gentle laser to the healthy nerve tissue. This laser treatment, known as "biomodulation," is thought to help calm the tissue and improve healing.

Patients who join the study will be randomly assigned to one of these two treatment groups. The main thing we will measure is the level of pain after the procedure, which patients will record on a simple pain scale. We want to find out if using the laser in addition to the filling material leads to less pain and a better experience after the treatment.

This study will help dentists understand if combining this new sealing material with laser therapy can be a more effective and comfortable way to save a tooth with a severe toothache.

DETAILED DESCRIPTION:
This study is a prospective, triple-blind, randomized controlled trial with two parallel arms and a 1:1 allocation ratio. It investigates the efficacy of adjunctive Er,Cr:YSGG laser biomodulation in managing postoperative pain following full pulpotomy procedures in permanent molars diagnosed with symptomatic irreversible pulpitis.

The standard of care for teeth with this diagnosis has traditionally been non-surgical root canal treatment (NSRCT), which involves the complete removal of the dental pulp. However, with the advent of advanced bioceramic materials like calcium silicate cements, Vital Pulp Therapy (VPT), specifically pulpotomy, has emerged as a scientifically valid treatment alternative for mature permanent teeth. Pulpotomy aims to preserve the vitality and health of the radicular pulp tissue, potentially offering biological advantages such as maintaining the tooth's proprioceptive and defensive mechanisms, while also being a less complex and more time-efficient procedure.

The primary material under investigation is EndoCem, a premixed, ready-to-use calcium silicate cement. These materials are favored in VPT due to their excellent bioactivity, biocompatibility, and ability to form a hermetic seal over the vital pulp tissue. The experimental intervention involves the application of Er,Cr:YSGG laser energy to the exposed radicular pulp stumps following hemostasis, prior to the placement of the EndoCem cement. The laser parameters will be set to a non-ablative, bio-stimulatory mode. The proposed mechanism of action includes biostimulation of pulpal fibroblasts and stem cells, enhanced local microcirculation, and anti-inflammatory effects, which collectively may lead to a more favorable and less painful postoperative healing response.

Participants will be recruited from the patient pool presenting at the outpatient clinic. After screening against the eligibility criteria, eligible participants (or their guardians) who provide informed consent will be randomized into one of two groups:

Group 1 (Control): Will receive a full pulpotomy procedure followed by the application of EndoCem cement as the pulpal medicament and final restoration.

Group 2 (Intervention): Will receive an identical full pulpotomy procedure, followed by Er,Cr:YSGG laser biomodulation of the pulp stumps, and then the application of EndoCem cement and final restoration.

The randomization sequence will be computer-generated, and allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes. To maintain blinding, the operating clinician will not be involved in postoperative assessments. The participant, the outcome assessor (who collects the pain scores), and the statistician analyzing the data will all be blinded to the group assignments.

The primary outcome is postoperative pain, which will be quantitatively measured using a Visual Analogue Scale (VAS). Participants will record their pain levels at predetermined time points following the procedure (e.g., 6, 12, 24, and 48 hours). The data will be analyzed to compare the mean pain scores and the incidence of moderate-to-severe pain between the two groups over time.

This study aims to provide high-level evidence on the potential synergistic effect of laser biomodulation when combined with modern bioceramics in VPT. The results could contribute to optimizing clinical protocols for managing irreversible pulpitis, shifting the paradigm towards more conservative, pulp-preserving treatments that enhance postoperative patient comfort.

ELIGIBILITY:
Inclusion Criteria:

Patients between 9 and 14 years of age. Must have a two-rooted mandibular molar tooth (lower back tooth). The tooth must be diagnosed with symptomatic irreversible pulpitis (a painful, inflamed nerve).

The tooth must be considered restorable (can be fixed with a filling or crown). Patient and/or guardian must be able to understand and sign the informed consent form.

The tooth must be periodontally healthy, with no mobility, and not painful to tapping or pressing.

Exclusion Criteria:

Teeth with immature root tips. Teeth that are not restorable (severely damaged or decayed). Bleeding from the tooth's nerve that cannot be controlled within 10 minutes during the procedure.

Patients with significant medical conditions that could complicate dental treatment.

Teeth with a dead (necrotic) nerve. Inability or unwillingness to provide informed consent. Individuals from vulnerable groups (as defined by the ethics committee).

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity as assessed by Visual Analogue Scale (VAS) | At 6, 12, 24, and 48 hours after the completion of the pulpotomy procedure.
  Postoperative pain level will be self-reported by participants using a 100-mm Visual Analogue Scale (VAS). The scale is a horizontal line anchored by two verbal descriptors: "No pain" (0 mm) on the left and "Worst pain imaginable" (100 mm) on the right. Participants mark the line at the point that best represents their pain intensity. A higher score indicates greater pain. The outcome for analysis is the mean VAS score recorded at each specified postoperative time point.

SECONDARY OUTCOMES:
Clinical Success Rate | At 1 week and 6 months post-treatment.
  The absence of clinical signs and symptoms of failure, including spontaneous pain, pain on palpation, pain on percussion, soft tissue swelling, sinus tract, or pathological tooth mobility. The outcome is reported as the number of participants with a clinically successful outcome.
Radiographic Success Rate | At 6 months post-treatment.
  The absence of radiographic signs of failure, assessed via periapical radiographs. This includes the absence of new or enlarged periapical radiolucency, external or internal root resorption, or periodontal ligament space widening. The outcome is reported as the number of participants with a radiographically successful outcome.

OTHER OUTCOMES:
Incidence of Analgesic Medication Use | Within 48 hours after the completion of the pulpotomy procedure.
  The number of participants who take rescue analgesic medication (e.g., Ibuprofen) for pain relief following the procedure. This is used as an indirect, patient-driven measure of significant postoperative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Medhat Kataia, PhD, Principal Investigator — Fujairah University
Locations (1):
- Dental Clinic, College of Dentistry, Fujairah University, Fujairah, Emirate of Fujairah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanna SN, Perez Alfayate R, Prichard J. Vital Pulp Therapy an Insight Over the Available Literature and Future Expectations. Eur Endod J. 2020 Mar 1;5(1):46-53. doi: 10.14744/eej.2019.44154. eCollection 2020. PMID 32342038
- [Background] Kim M, Yang W, Kim H, Ko H. Comparison of the biological properties of ProRoot MTA, OrthoMTA, and Endocem MTA cements. J Endod. 2014 Oct;40(10):1649-53. doi: 10.1016/j.joen.2014.04.013. Epub 2014 Jul 19. PMID 25052144
- [Background] Kaur M, Singh H, Dhillon JS, Batra M, Saini M. MTA versus Biodentine: Review of Literature with a Comparative Analysis. J Clin Diagn Res. 2017 Aug;11(8):ZG01-ZG05. doi: 10.7860/JCDR/2017/25840.10374. Epub 2017 Aug 1. PMID 28969295
- [Background] Drouri S, El Merini H, Sy A, Jabri M. Evaluation of Direct and Indirect Pulp Capping With Biodentine in Vital Permanent Teeth With Deep Caries Lesions. Cureus. 2023 May 23;15(5):e39374. doi: 10.7759/cureus.39374. eCollection 2023 May. PMID 37250608
- [Background] Stanley HR. Pulp capping: conserving the dental pulp--can it be done? Is it worth it? Oral Surg Oral Med Oral Pathol. 1989 Nov;68(5):628-39. doi: 10.1016/0030-4220(89)90252-1. PMID 2682429
- [Background] Caplan DJ, Cai J, Yin G, White BA. Root canal filled versus non-root canal filled teeth: a retrospective comparison of survival times. J Public Health Dent. 2005 Spring;65(2):90-6. doi: 10.1111/j.1752-7325.2005.tb02792.x. PMID 15929546
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Background] Rebel, H-H. (1922). "über die Ausheilung der freigelegten pulpa". Ditsch Zahnheilkd.